CLINICAL TRIAL: NCT06425640
Title: INTERPLAY WITHIN THE DAY: Optimizing Intra-day Glucose Control by Intervening on the Day-to-day 24-hour Movement Behavior Patterns in Adults With Type 1 Diabetes Mellitus.
Brief Title: 24-hour Movement Behaviors in Adults With Type 1 Diabetes
Acronym: 24h-MBs_T1D
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2023-0611
Record Dates: First submitted 2024-05-01; First posted 2024-05-22 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: 24-hour movement behaviors; Glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with type 1 diabetes: Adults with type 1 diabetes (25-50 years) will wear an accelerometer to objectively measure their 24-hour movement behaviors. An online questionnaire and food diary will be completed to gain insight into the explanatory variables of 24-hour movement behaviors. Information on glucose control will be collect through the continuous glucose monitor of the participant.
  Interventions: Behavioral: 24-hour movement behavior

INTERVENTIONS:
Behavioral: 24-hour movement behavior — Cross-sectional observational study investigating the 24-hour movement behaviors and glucose control

SUMMARY:
Only 24.9% of the Belgian adults (25-50 years) with type 1 diabetes mellitus (T1DM) achieve a good glucose control. This can be explained by the challenging day-to-day diabetes management which places a substantial burden on this population. However, a tight glycemic control is fundamental in order to prevent the development of acute and chronic complications. Despite the added value of continue glucose monitors to glucose control, optimizing daily glucose levels is still problematic in adults with T1DM. In addition to self-monitoring of blood glucose, a healthy lifestyle with sufficient physical activity (PA), limited sedentary behavior (SB) and sufficient sleep time and quality is crucial for a good glucose control. A recent shift in health promotion stresses the importance of considering all these behaviors (i.e. PA, SB and sleep) in one 24-hour day instead of focusing on one behavior in isolation. The aim of this study is to investigate the association between the day-by-day 24h-MB patterns of adults (25-50 years) with T1DM and their intra-day glucose control (i.e. time in range and coefficient of variation) on the one hand. On the other hand, associations between he 24-h MB patterns and explanatory variables and cardiometabolic health markers will be investigated. To gain insight into the 24-hour behavior of adults with type 1 diabetes, 150 adults with type 1 diabetes will wear an Actigraph accelerometer, for 14 consecutive days. Daily glucose control will be measured using the participant's continuous glucose meter. Information about the explanatory variables and cardiometabolic health will be obtained by means of a questionnaire, diary and a few measurements (blood pressure, weight, length, Advanced Glycation Endproducts, hip-and waist circumference) during a one-off visit to one of the recruitment- and testing centers namely University hospital of Ghent or University hospital of Antwerp. The results of this cross-sectional study will inform future interventions focusing on the 24-hour movement behaviors in adults with T1DM.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 25 and 50 years
* Diagnosed with T1DM for a minimum of two years
* Minimal daily insulin dose of 10 units
* Using a continuous glucose monitor
* Most recent HbA1c between 6% and 9.5%

Exclusion Criteria:

* Using a hybrid closed loop insulin pump
* Shift workers
* Known cardiovascular disease (e.g. peripheral arterial disease causing intermittent claudication reducing walking distance to <500 meters, history of cerebrovascular accidents with residual impact on motoric function or heart failure NYHA class 3 and 4)
* Physical disabilities that disturb daily functioning (e.g. amputations, paralysis)
* Other conditions affecting normal movement behaviors (e.g. active treatment for malignancies, diabetic nephropathy stage 4 or 5, chronic obstructive pulmonary disease stage 3 or 4 or asthma stage 3 or 4)
* Visual impairment (e.g. retinopathy with loss of vision or blindness)
* Hypoglycemia unawareness (i.e. self-reporting of biochemical hypoglycemia unaccompanied by symptoms, loss of autonomic symptoms (e.g. hunger, sweating) as initial sign of hypoglycemia)
* Symptomatic peripheral neuropathy(i.e. loss of sensations, pain, exaggerated sensitivity to painless stimuli, paresthesia, ulceration injuries or amputations)
* Professional or semi-professional top athletes
* Participating in another supervised healthy lifestyle or drug intervention

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A total of 150 adults (25-50 years) with T1DM will be recruited in this study. Participants will be recruited through visits at diabetologists at University hospital of Ghent and Antwerp, diabetes educators, dieticians, general practitioners and community health centres.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
24-hour movement behaviors | Through study completion, an average 1 year
  All the movement behaviors performed within one day (i.e. PA, SB and sleep) will be objectively measured using an Actigraph wGT3X-BT accelerometer. The participants will wear the accelerometer for 14 consecutive days. At daytime, the accelerometer will be worn at the right hip, at night the accelerometer will be switched to the non-dominant wrist.
Coefficient of variation (in %) | Through study completion, an average 1 year
  Coefficient of variation is a measure for intra-day glucose control and will be measured by the continuous glucose monitor of the participants. Raw CGM data of 14 consecutive days will be downloaded from the receiver of the participants with the programme compatible with their CGM (i.e. Libreview, Dexcom studio, Glooko).
Time in range | Through study completion, an average 1 year
  Time in range is a measure for intra-day glucose control and will be measured by the continuous glucose monitor of the participants. Raw CGM data of 14 consecutive days will be downloaded from the receiver of the participants with the programme compatible with their CGM (i.e. Libreview, Dexcom studio, Glooko).

SECONDARY OUTCOMES:
Waist circumference (in cm) | Through study completion, an average 1 year
  Waist circumference will be measured twice with a measuring tape (Seca 201).
Hip circumference (in cm) | Through study completion, an average 1 year
  Hip circumference will be measured twice with a measuring tape (Seca 201).
Blood pressure (in mmHg) | Through study completion, an average 1 year
  Blood pressure will be measured twice with an interval of one minute with an automatic OMRON M6 Comfort device after 10 minutes of rest.
Advanced glycation endproducts | Through study completion, an average 1 year
  AGE's, a predictive value for the development of diabetic and cardiovascular complications, will be measured with a skin AGE-reader (Diagnoptics Technologies, Groningen, the Netherlands).
LDL-cholesterol (in mg/dl) | Through study completion, an average 1 year
  LDL-cholesterol will be obtained through the participants' most recent blood results.
HDL-cholesterol (in mg/dl) | Through study completion, an average 1 year
  HDL-cholesterol will be obtained through the participants' most recent blood results.
Triglycerides (in mg/dl) | Through study completion, an average 1 year
  Triglycerides will be obtained through the participants' most recent blood results.
Total cholesterol (in mg/dl) | Through study completion, an average 1 year
  Total cholesterol will be obtained through the participants' most recent blood results.
Long-term glucose regulation (in % or mmol/mol) | Through study completion, an average 1 year
  Average HbA1c over the last 10 years (or from diagnosis if diagnosis was less than 10 years ago) will be collected through the patient file.
Medication intake | Through study completion, an average 1 year
  Information about medication intake will be collected through the patient file.
C-peptide level | Through study completion, an average 1 year
  Information about C-peptide level will be collected through the patient file.
Co-morbidities | Through study completion, an average 1 year
  Information about comorbidities will be collected through the patient file.
Weight (in kg) | Through study completion, an average 1 year
  Weight will be collected through the patient file.
Mean glucose | Through study completion, an average 1 year
  The mean glucose of 14 consecutive days will be derived from the participant's raw CGM data.
Standard deviation | Through study completion, an average 1 year
  The standard deviation of glucose, a measure of the spread in glucose readings around the average glucose, will be derived from the participant's raw CGM data.
Mean amplitude of glycemic excursions | Through study completion, an average 1 year
  Mean amplitude of glycemic excursions, a glucose variability metric, will be derived from the participant's raw CGM data.
Continuous overall net glycemic action | Through study completion, an average 1 year
  Continuous overall net glycemic action, a measure of glycemic variability, will be derived from the participant's raw CGM data.
Percent of measurements below 70 mg/dl (in %) | Through study completion, an average 1 year
  Percent of measurements below 70 mg/dl, a measure that gives insight in the time in hypoglycemia, will be derived from the participant's raw CGM data.
Percent of measurements above 180 mg/dl (in %) | Through study completion, an average 1 year
  Percent of measurements above 180 mg/dl, a measure that gives insight in the time in hyperglycemia, will be derived from the participant's raw CGM data.
Mean of daily differences | Through study completion, an average 1 year
  Mean of daily differences, a measure that gives insight in the between-days glycemic variability, will be derived from the participant's raw CGM data.

OTHER OUTCOMES:
Demographics | Through study completion, an average 1 year
  Following demographics will be questioned in a self-developed questionnaire: age, sex, ethnicity, smoking status, educational level, profession, family situation.
Health-related variables | Through study completion, an average 1 year
  Health-related variables that will be questioned are height, weight, timing of T1DM diagnosis, insulin delivery system (CSII versus multiple daily injections), insulin and other medication.
Health-related quality of life | Through study completion, an average 1 year
  Two questionnaires will be used to measure HRQOL: the Short Form 36 health survey questionnaire (SF-36) and the Diabetes Quality of life questionnaire-brief (DQOLQ-brief). The SF-36 will measure the general HLQOL. The DQOLQ-brief will assesses diabetes-related QOL.
Depression an anxiety | Through study completion, an average 1 year
  The Hospital Anxiety and Depression Scale is a short (14-item) and easy to use questionnaire. The questionnaire consists of two subscales: one evaluates anxiety (7 items) and the other depression (7 items).
Diabetes knowledge | Through study completion, an average 1 year
  The patient education and knowledge (PEAK) questionnaire will be used to assess diabetes knowledge. Diabetes knowledge is determined based on 10-items (i.e. knowledge about insulin titration, correction factor, carbohydrate counting, PA and interpretation of glucose trends) with scores ranging from 0 (no diabetes knowledge) to 10 (excellent diabetes knowledge).
Health literacy | Through study completion, an average 1 year
  Health literacy will be assessed using the validated Newest-Vital Sign-D (NVS-D) questionnaire. The NVS-D is a six items questionnaire which assesses an individual ability to find, understand and apply information.
Diabetes self-management | Through study completion, an average 1 year
  Diabetes self-management will be assessed using the diabetes self-management questionnaire revised (DSMQ-R). The DSMQ-R is a multidimensional validated questionnaire with 27-items regarding essential self-management practices (e.g. glucose monitoring, physical activity, cooperation with diabetes team) for T1DM.
Behavioral factors | Through study completion, an average 1 year
  newly developed and reliable questionnaire to assess explanatory variables 24h-MBs in adults will collect information on behavioral factors. The behavioral factors are based on the integrated behavior change (IBC) model. This model combines different behavioral change theories, i.e. the theory of planned behavior, the self-determination theory, and the dual system theory. The following behaviors will be questioned: autonomous motivation, attitude, internal behavioral control (i.e. habits, skills), external behavioral control (i.e. barriers) and self-efficacy. The validated barriers to physical activity in T1DM (BAPD-1) questionnaire will assess external behavioral control factors for physical activity.
Environmental factors | Through study completion, an average 1 year
  A newly developed and reliable questionnaire to assess explanatory variables of 24-h movement behaviors in adults will collect information on socio-environmental factors and physical environmental factors. The socio-environmental factors are subjective norm, social modelling and social support. The physical environmental factors are electronic devices at home, sleep environment, neighbourhood and work environment.
Context-related information about physical activity | Through study completion, an average 1 year
  Each accelerometer will be supplemented by a diary in which the participant will be asked to give context-related information about PA (e.g. type of sport, active transportation) and sleep (e.g. sleep quality).
Food intake | Through study completion, an average 1 year
  Dietary intake, an important and indispensable component of diabetes management, will be measured with a 14-day food diary completed during the same period of wearing the ActiGraph. Since a written food diary is time consuming and can result in reporting errors (i.e. underreporting due to difficulties in estimating portion sizes), the Digitaal Dagboek application (https://digitaaldagboek.be/) will be used to register daily food intake.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Lapauw, Professor, Principal Investigator — University Hospital, Ghent; Eveline Dirinck, Professor, Principal Investigator — University Hospital, Antwerp; Marieke De Craemer, Professor, Principal Investigator — University Ghent
Locations (2):
- Belgium (2):
  - University Hospital Ghent, Ghent, East Flanders
  - University Hospital Antwerp, Antwerp